CLINICAL TRIAL: NCT06451328
Title: Lignosus Rhinoceros TM02® as a Complementary Therapy for Uncontrolled Asthma: A Prospective, Open-label, Single-arm, Phase II Study
Brief Title: Lignosus Rhinoceros TM02® as a Complementary Therapy for Uncontrolled Asthma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Malaya (Other)
Responsible Party: Principal Investigator, Poh Mau Ern, Associate Professor Dr, University of Malaya
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202010239161
Record Dates: First submitted 2024-05-28; First posted 2024-06-11 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Asthma
Keywords: asthma; FeNO; FEV1; Lignosus rhinoceros; TM02®
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TM02® (Experimental): Two capsules of TM02®, once daily after meals (breakfast or dinner), totaling 600 mg TM02® daily for 30 days. Subsequently, two capsules of 300 mg TM02®, twice a day after breakfast and dinner daily, totaling 1200 mg TM02® daily for an additional 60 days.
  Interventions: Drug: Lignosus rhinoceros TM02®

INTERVENTIONS:
Drug: Lignosus rhinoceros TM02® — Lignosus rhinoceros TM02®

SUMMARY:
The goal of this clinical trial is to learn if TM02® works to treat partially controlled or uncontrolled asthma in adults. It will also learn about the efficacy and safety of TM02®.

The main questions it aims to answer are:

Does TM02® causes bronchodilation (to what extent), improves asthma control, and reduces airway inflammation and blood eosinophils and serum immunoglobulin E levels.

Participants will:

Take TM02® every day for 90 days. Visit the clinic once every 30 days for checkups, tests and to fill up questionnaires.

Keep a diary of their symptoms and the number of times they use a rescue inhaler.

DETAILED DESCRIPTION:
This 90-day prospective phase II, open label, single-arm study was conducted from March 2022 to February 2023. Subjects with partially controlled or uncontrolled asthma, assessed according to the Global Initiative for Asthma (GINA) guidelines, were enrolled from the outpatient asthma clinic at the Universiti Malaya Medical Centre, Kuala Lumpur, Malaysia. The effects of TM02® on bronchodilation was determined via trough forced expiratory volume in 1 second (FEV1) assessment. Improvement of asthma control was assessed using the Asthma Control Questionnaire-7 (ACQ-7). Serial measurements of fractional exhaled nitric oxide (FeNO) levels at baseline, 30, 60 and 90 days were performed to assess the effectiveness of TM02® in reducing FeNO, a marker of Type 2 airway inflammation. Blood eosinophil count and serum immunoglobulin E (IgE) level were also measured.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years and above with a prior documented diagnosis of asthma by a physician based on the GINA guidelines following these criteria: well-documented requirement for regular treatment with a minimum dose of either fluticasone/salmeterol combination therapy or budesonide/formoterol combination therapy for three months, with a stable dose for one month prior to screening, FEV1 >35% to <80% measured during the screening phase (3 attempts maximum) prior to the first dose of TM02®, reversibility of at least 12% and 200 mL in FEV1 after 400 mcg salbutamol during the screening phase, or documented history of reversibility test that met these criteria within 12 months prior to screening.
* No recent exacerbations six weeks prior to enrolment
* Non-smoker for at least one year with a prior tobacco consumption < 10 pack-years
* Normal organ function; and weigh > 41 kg with a body mass index (BMI) between 18 and 35 kg/m2.

Exclusion Criteria:

* Currently exposed to allergens or triggering factors influencing asthma control
* Pregnant or lactating
* Have chronic obstructive pulmonary disease (COPD) and/or other lung diseases impairing pulmonary function test
* Receiving oral corticosteroids for any other reason than to treat asthma within 6 weeks prior to screening
* Had history of acute sinus infection or respiratory tract infection within 4 weeks prior to screening
* Cardiac disorders which include one of the following conditions: acute coronary syndrome, acute heart failure [Class III or IV of the New York Heart Association (NYHA) classification], ventricular arrhythmia (persistent ventricular tachycardia, ventricular fibrillation, resuscitated sudden death), cardiac failure class III or IV of the NYHA classification, severe conduction disorders which are not prevented by permanent pacing (atrio-ventricular block 2 and 3, sino-atrial block), syncope with unknown etiology within 3 months, or uncontrolled hypertension.
* Active lung disease other than asthma (eg. chronic bronchitis)
* Had undergone major surgery within 4 weeks prior to screening
* Have a life expectancy of less than 6 months
* Had a history of primary malignancy < 5 years (except treated basal cell skin cancer or cervical carcinoma in situ)
* Had any severe and/or uncontrolled medical condition aside from asthma
* Has human immunodeficiency virus (HIV) infection
* Had a history of poor compliance or drug/alcohol abuse,
* Had participated in a clinical study with exposure to any non-registered drug or botanical product within 30 days prior
* Had a condition that would interfere with their ability to provide informed consent, comply with the study protocol, or put the person in undue risk.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Changes in mean trough FEV1 in millilitres from baseline (pre-treatment) to end of the 90-day treatment period | 90 days
  Mean trough FEV1 in millilitres
Mean change in Asthma Control Questionnaire -7 (ACQ - 7) scores from baseline (pre-treatment) to end of the 90-day treatment period | 90 days
  The ACQ-7 consists of 6 questions about asthma symptoms during the previous week, each of which is scored on a range from 0 (no impairment) to 6 (maximum impairment), and an assessment of FEV1. The minimal clinically important difference (MCID) is 0.5 units.

SECONDARY OUTCOMES:
Changes in mean FeNO levels in parts per billion (ppb) from baseline to end of the 90-day treatment period | 90 days
  Mean FeNO in parts per billion (ppb)
Changes in mean blood eosinophil count in cells per decilitre (cells/dL) from baseline to end of the 90-day treatment period | 90 days
  Mean blood eosinophil count in cells per decilitre
Changes in mean serum immunoglobulin E level in International units per millilitre (IU/ml) from baseline (pre-treatment) to end of the 90-day treatment period. | 90 days
  Mean serum immunoglobulin E level in International unit per millilitre (IU/ml)

CONTACTS AND LOCATIONS:
Overall Officials: Mau Ern Poh, MBBS, Principal Investigator — Universiti Malaya
Locations (1):
- University of Malaya Medical Centre, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2021-02-14): https://cdn.clinicaltrials.gov/large-docs/28/NCT06451328/Prot_000.pdf
  • Informed Consent Form (2020-10-23): https://cdn.clinicaltrials.gov/large-docs/28/NCT06451328/ICF_001.pdf